CLINICAL TRIAL: NCT03254563
Title: Copeptin and Nonalcoholic Fatty Liver Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 17-1160
Record Dates: First submitted 2017-08-16; First posted 2017-08-18 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum and urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Obese with NAFLD: Patients who have NAFLD based upon ultrasound
- Obese without NAFLD: Patients who do not have NAFLD based upon ultrasound

SUMMARY:
Copeptin, a surrogate marker for vasopressin, has been found to be elevated in metabolic disorders including obesity and diabetes, which are disorders both associated with nonalcoholic fatty liver disease (NAFLD), and therefore suggest a potential role for vasopressin in the pathogenesis of NAFLD. The investigators intend to investigate if there is an association of vasopressin with the presence and severity of NAFLD.

DETAILED DESCRIPTION:
Participants: As a pilot study, the investigators will recruit 30 obese adults with NAFLD based upon ultrasound echogenicity within 6 months of enrollment, and 30 obese adults without NAFLD based upon ultrasound (US) echogenicity for comparison.

Screening Visit/Study Visit: Patients in the investigator's Obesity clinic will be approached about the study and consented if interested at the screening. Participants will have a chart review for their history and physical Exam and medication review for inclusion and exclusion criteria. Qualified participants will be invited for a screening visit to be scheduled in conjunction with the labs and procedures performed as Standard of Care (SOC) in the obesity clinic. At the screening visit, following consent, participants will have vitals (blood pressure, Body Mass Index (BMI), waist circumference) and a physical examination performed. Participants' Standard of Care (SOC) labs including fasting lipid panel, HbA1c (unless done within last 3 months), comprehensive metabolic panel, titers for hepatitis b and c, and complete blood count will be drawn, along with the following research labs: insulin, glucagon, free fatty acids, adiponectin and a 24-hour urine cortisol collection. Those who have not had an abdominal US will have a SOC US performed to delineate non-NAFLD or NAFLD status. US will not be performed if already done within 6 months of enrollment. All ultrasound studies will be interpreted by one University of Colorado Denver radiologist to categorize the patient as NAFLD or non-NAFLD to limit inter-reader variability. Those with NAFLD present on US will also have a SOC Fibroscan done to assess severity of steatosis (based upon Controlled Attenuation Parameter or CAP Score) and fibrosis (based upon elastography). Given limitations of ultrasound to accurately detect significant steatosis unless >30%, the investigators will in addition perform Fibroscan (all particpants regardless of US) to assess steatosis, so as to confirm if significant steatosis and compare copeptin levels on a continuum of level of steatosis as part of research procedure. Fibroscan can detect steatosis (based upon Controlled Attenuation Parameter or CAP Score) and fibrosis (based upon elastography). FIbroscan with M probe has been found to have AUROC 0.823 for a cutoff of value of 248 dB/m for no steatosis vs steatosis (with other cutoffs at 268 dB/m between S1 and S2-S3 and 280 dB/m between S1-S2 and S3 disease).

ELIGIBILITY:
Inclusion Criteria:

1. Patients age 30-75
2. BMI 30-40
3. Presence of fatty liver on ultrasound

Exclusion Criteria:

1. Diabetes mellitus (determined by prior HbA1c, fasting glucose, and/or random glucose in the last three months according to ADA criteria),
2. Medication known to affect insulin sensitivity e.g. metformin, thiazolidinediones, systemic steroids, atypical antipsychotics),
3. Fibrates,
4. eGFR <45 ml/min/1.73m2 by MDRD equation(11),
5. Pregnancy,
6. Breast feeding,
7. Sodium <135 mEq/L,
8. Diabetes insipidus,
9. Liver disease other than NAFLD (including obstructive liver disease),
10. ALT or AST>60 IU/L,
11. Hepatic steatosis on ultrasound for the non-NAFLD group,
12. Congestive heart failure,
13. Patients who consume >20g of ETOH a day,
14. Patients found to have Cushing's disease based upon 24 hour urine results (Urine Free cortisol >2x upper limit of normal).
15. Patient's with pacemakers
16. Off of Coenzyme Q for 6 months.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Obese adults (BMI 30-40 kg/m2) age 30-75 years with NAFLD based upon ultrasound echogenicity within 6 months of enrollment
  2. Obese adults (BMI 30-40 kg/m2) age 30-75 years without NAFLD based upon ultrasound echogenicity within 6 months of enrollment
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-06-19 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Comparision of Copeptin with and without NAFLD | Within 6 months of documented NAFLD or non-NAFLD and within 1 week of fibroscan
  The investigators will compare level of copeptin with the measurement of NAFLD based upon ultrasound and fibroscan.
Copeptin and level of steatosis | Within one week of fibroscan being perfomed
  Comparison of CAP score of fibroscan to copeptin levels
Copeptin and Liver Elastography | Within one week of fibroscan being perfomed
  Compare Copeptin to liver elastography (kPa)

SECONDARY OUTCOMES:
Insulin Resistance and copeptin | Same day as these labs after 8 hour fast from food and water.
  Changes in insulin, fasting glucose, HOMA-IR, HOMA-B, adiponectin estimated Insulin Compared to copeptin level
Copeptin and Lipids | Same day as these labs after 8 hour fast from food and water.
  Compare copeptin level to cholesterol and free fatty acids
Copeptin and Liver enzymes | Same day as these labs after 8 hour fast from food and water.
  Compare copeptin and liver enzymes
Copeptin and Weight | Within 1 month of screening visit
  Compare Copeptin with BMI
Copeptin and Waist Circumference | Within 1 month of screening visit
  Compare copeptin with weight circumference
Copeptin and Blood pressure | Within 1 month of screening visit
  Compare copetin with measurements of blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Jensen, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No